CLINICAL TRIAL: NCT00974636
Title: Lowering Salt Intake in Chronic Kidney Disease: A Pilot Randomized Crossover Trial
Acronym: BIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Renal Research Institute (Other)
Responsible Party: Principal Investigator, Rajiv Saran, MD, MS, MRCP, Associate Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: HUM00016384
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Kidney Disease
Keywords: Kidney Disease; Albuminuria; Glomerular filtration rate; Volume status; Bioimpedance analysis
MeSH Terms: conditions — Kidney Diseases; Albuminuria | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Salt Diet (Experimental): Dietary sodium restriction of ≤2.0 g/day or ≤ 85 mmol/day for two weeks
  Interventions: Dietary Supplement: Low Salt Diet
- Ususal Salt Diet (Placebo Comparator): Usual salt intake (approximately >180-200 mmol/day in the average American diet).
  Interventions: Dietary Supplement: Usual Salt Diet

INTERVENTIONS:
Dietary Supplement: Low Salt Diet — Dietary sodium restriction of ≤2.0 g/day or ≤ 85 mmol/day
  Other Names: Low salt diet, CKD, Bioimpedance analysis (BIA)
  Arms: Low Salt Diet
Dietary Supplement: Usual Salt Diet — Usual salt intake (approximately >180-200 mmol/day in the average American diet).
  Arms: Ususal Salt Diet

SUMMARY:
ABSTRACT

Background:

It is well recognized that excess dietary salt intake plays a major role in the development of hypertension. Chronic Kidney Disease (CKD) is associated with excess salt and water retention (excess volume) which is associated with hypertension.

Hypotheses:

Hypothesis 1:

Dietary salt restriction will improve volume status in subjects with CKD stages 3-4 as assessed by Bioelectrical Impedance Analysis (BIA).

Hypothesis 2:

Dietary salt restriction will result in improved blood pressure control in patients with CKD stages 3-4.

Hypothesis 3:

Dietary salt restriction will decrease albuminuria in patients with CKD stages 3-4.

Patients and Trial Design: This randomized crossover pilot study is designed to assess the effect of salt restriction on volume status in patients with CKD stages 3 and 4.

Subjects will be randomized to a treatment order: (1) 4 weeks of salt restriction of <85 mmol sodium per day, a 2 week washout period, and 4 weeks of usual salt diet, OR (2) 4 weeks of usual diet, 2 weeks washout, and 4 weeks of salt restriction. Patients will receive dietary counseling in person at each study visit and at weekly intervals by phone calls from study dieticians. At weeks 0, 4, 6 and 10, patients will undergo assessments for (i) physical examination with assessments for weight, blood pressure, pulse, anthropometrics and a standardized clinical assessment of volume status. (ii) volume status using bioelectrical impedance analysis (BIA) (iii) 24-hour urine testing for, albumin, creatinine and aldosterone Every 2 weeks throughout the study, a 24-hour urine sodium will be measured for compliance, and serum electrolytes will be assessed for safety.

Data Analysis: BIA measurements in the low salt group will be compared with the regular diet group using the standard linear model analysis for 2x2 crossover trials. Additionally, 24-hour ambulatory and static blood pressure and 24-hour urine aldosterone levels will be compared between the two groups.

Future Implications: A significant reduction in the degree of volume expansion (as assessed by BIA) and blood pressure as a result of a salt restricted diet would have implications for renal and cardiovascular protection and would warrant confirmation by a larger randomized trial.

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible to participate in this study must meet all of the following criteria:

* Willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures.
* Age ≥ 18 years and ≤ 85 years.
* Willing and able to comply with all study procedures.
* Patients with eGFR of 20 to 60 ml/min/173m2 by the abbreviated (4-variable) MDRD equation and a relatively stable clinical course.
* Sitting systolic blood pressure ≥ 100 mmHg prior to study entry (to exclude people at risk from hypotension from dietary salt reduction).

Exclusion Criteria:

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

* Recent acute illness (≤1 month). Minor ailments such as a recovered common cold or allergic rhinitis would not be considered as exclusion criteria but would be left to the site PI's discretion.
* Recent hospitalization (≤1 month) unless clearly for a minor elective procedure unlikely to interfere with BIA measurements. The final decision will be left to the site PI's discretion.
* Any psychological condition (including alcoholism) that could interfere with the patient's ability to comply with the study protocol.
* Subjects with baseline 24-hour urinary sodium excretion ≤100 mmol/day.
* Amputation of a limb other than fingers or toes.
* Pacemaker, defibrillator, implantable pump, artificial joint, pins, plates or other types of metal objects in the body (other than dental fillings).
* Coronary stents or metal suture material in the heart.
* Use of any investigational product or investigational medical device within 30 days prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
* Weight over 300 pounds (limitation for examination table).
* Pregnancy or lactation.
* Patients with kidney diseases known to be associated with salt wasting (see above).
* Patients with atrial fibrillation as ambulatory blood pressure measurements may not be accurate in this setting.
* Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-05; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Primary Outcome: Change in volume status (intracellular, extracellular volume, and total body water) as measured by BIA using both whole body and segmental techniques | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Saran, MD, Principal Investigator — University of Michigan
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] McMahon EJ, Campbell KL, Bauer JD, Mudge DW, Kelly JT. Altered dietary salt intake for people with chronic kidney disease. Cochrane Database Syst Rev. 2021 Jun 24;6(6):CD010070. doi: 10.1002/14651858.CD010070.pub3. PMID 34164803